CLINICAL TRIAL: NCT03320941
Title: A Randomized, Double-blind, Dose-finding Study to Evaluate the Change in Weight After 12 Weeks Treatment With 4 Doses of LIK066 Compared to Placebo in Japanese Patients With Obesity Disease
Brief Title: A Dose-finding Study to Evaluate the Change in Weight After Treatment With LIK066 in Japanese Patients With Obesity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CLIK066B1201
Record Dates: First submitted 2017-10-22; First posted 2017-10-25 (Actual); Results first posted 2019-10-02 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Obesity
Keywords: Obesity disease; Over weight; T2DM; interventional study; Weight loss
MeSH Terms: conditions — Obesity; Weight Loss | interventions — licogliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Parallel Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- LIK066 2.5 mg (Experimental): Eligible patients randomized to this arm will receive LIK066 2.5 mg orally daily for 12 weeks.
  Interventions: Drug: LIK066
- LIK066 10 mg (Experimental): Eligible patients randomized to this arm will receive LIK066 10 mg orally daily for 12 weeks.
  Interventions: Drug: LIK066
- LIK066 25 mg (Experimental): Eligible patients randomized to this arm will receive LIK066 25 mg orally daily for 12 weeks.
  Interventions: Drug: LIK066
- LIK066 50 mg (Experimental): Eligible patients randomized to this arm will receive LIK066 50 mg orally daily for 12 weeks.
  Interventions: Drug: LIK066
- Placebo (Placebo Comparator): Eligible patient randomized to this arm will receive LIK066 matching placebo orally daily for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LIK066 — LIK066 will be supplied in different doses as tablets to be taken orally daily.
  Arms: LIK066 10 mg; LIK066 2.5 mg; LIK066 25 mg; LIK066 50 mg
Drug: Placebo — Placebo will be supplied as tablets to be taken daily orally.
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate the efficacy, tolerability and safety of LIK066 to support dose selection for Phase 3 development in Japanese adults with obesity disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients with obesity disease and inadequately controlled body weight with diet and/or exercise
* BMI ≥ 25 kg/m^2 combined with at least two obesity-related comorbidities, or BMI ≥ 35 kg/m^2 at least one obesity-related comorbidity
* Patients with FPG ≥ 110 mg/dL and/or 5.6% ≤ HbA1c ≤ 10.0%, or T2DM with HbA1c ≤ 10.0%
* Waist circumference at umbilical level ≥ 85 cm for male, ≥ 90 cm for female
* Visceral fat area ≥ 100 cm^2
* Agreement to comply with the study-required life-style intervention and treatment during the full duration of the study

Exclusion Criteria:

* Pregnancy or lactating women
* Use of pharmacologically active weight-loss medications
* Bariatric surgery
* Ketoacidosis, lactic acidosis, hyperosmolar coma
* Symptomatic genital ingection or urinary tract infection in the 4 weeks prior to screening
* Gastro-intestinal (GI) disorders associated with chronic diarrhea
* Congestive heart failure, New York Heart Association (NYHA) class III or IV

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2017-12-07 (Actual); Primary Completion 2018-07-25 (Actual); Study Completion 2018-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (19):
- Japan (19):
  - Novartis Investigative Site, Matsudo, Chiba
  - Novartis Investigative Site, Chikushino-shi, Fukuoka
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Kitakyushu, Fukuoka
  - Novartis Investigative Site, Akashi, Hyōgo
  - Novartis Investigative Site, Kakogawa, Hyōgo
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Kumamoto, Kumamoto
  - Novartis Investigative Site, Kyoto, Kyoto
  - Novartis Investigative Site, Nagasaki, Nagasaki
  - Novartis Investigative Site, Higashiosaka, Osaka
  - Novartis Investigative Site, Ageo, Saitama
  - Novartis Investigative Site, Kawaguchi, Saitama
  - Novartis Investigative Site, Tokorozawa, Saitama
  - Novartis Investigative Site, Hachiōji, Tokyo
  - Novartis Investigative Site, Kiyose, Tokyo
  - Novartis Investigative Site, Minato-ku, Tokyo
  - Novartis Investigative Site, Shinagawa-ku, Tokyo
  - Novartis Investigative Site, Toshima-ku, Tokyo

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Yokote K, Sano M, Tsumiyama I, Keefe D. Dose-dependent reduction in body weight with LIK066 (licogliflozin) treatment in Japanese patients with obesity. Diabetes Obes Metab. 2020 Jul;22(7):1102-1110. doi: 10.1111/dom.14006. Epub 2020 Mar 12. PMID 32072763
- See also: A Plain Language Trial Summary is available on novartisclinicatrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=432

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 126 participants were randomized and received at least one dose of study drug.
Groups:
- LIK066 2.5mg qd: Eligible patients randomized to this arm will receive LIK066 2.5 mg orally daily (qd) for 12 weeks.
- LIK066 10mg qd: Eligible patients randomized to this arm will receive LIK066 10 mg orally daily (qd) for 12 weeks.
- LIK066 25 mg qd: Eligible patients randomized to this arm will receive LIK066 25 mg orally daily (qd) for 12 weeks.
- LIK066 50 mg qd: Eligible patients randomized to this arm will receive LIK066 50 mg orally daily (qd) for 12 weeks.
Period: Overall Study
Arm/Group | LIK066 2.5mg qd | LIK066 10mg qd | LIK066 25 mg qd | LIK066 50 mg qd | Placebo
Started | 19 | 19 | 28 | 31 | 29
Completed | 19 | 19 | 28 | 30 | 29
Not Completed | 0 | 0 | 0 | 1 | 0
Not completed — subject/guardian decision | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LIK066 2.5mg qd | LIK066 10mg qd | LIK066 25 mg qd | LIK066 50 mg qd | Placebo | Total
Number analyzed (Participants) | 19 | 19 | 28 | 31 | 29 | 126
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.2 (10.44) | 57.2 (7.54) | 56.8 (9.50) | 57.9 (11.37) | 59.3 (9.76) | 57.7 (9.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 11 | 14 | 12 | 48
  Male | 15 | 12 | 17 | 17 | 17 | 78
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 19 | 19 | 28 | 31 | 29 | 126
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change From Baseline in Body Weight at Week 12
Description: The dose-response relationship of LIK066 as measured by percent change from baseline in body weight relative to placebo after 12 weeks of treatment.
Time Frame: Baseline, Week 12
Population: Full analysis set (FAS) - includes all 126 randomized participants that took at least one dose of study drug
Measure: Number (95% Confidence Interval); unit: Percent Change
Arm/Group | LIK066 2.5mg qd | LIK066 10mg qd | LIK066 25 mg qd | LIK066 50 mg qd | Placebo
Number analyzed (Participants) | 19 | 19 | 28 | 31 | 29
Percent Change | -1.86 [-2.59 to -0.67] | -2.84 [-3.79 to -2.16] | -3.41 [-3.96 to -2.84] | -3.80 [-4.48 to -3.17] | 0.11 [-0.90 to 0.97]
Statistical Analysis 1: Comparison: LIK066 2.5mg qd vs Placebo; Test type: Other — Dose Finding; Mean Difference (Net) = -1.99, 95% CI 2-sided [-2.92 to -0.21]
Statistical Analysis 2: Comparison: LIK066 10mg qd vs Placebo; Test type: Other — Dose Finding; Mean Difference (Net) = -3.00, 95% CI 2-sided [-4.15 to -1.70]
Statistical Analysis 3: Comparison: LIK066 25 mg qd vs Placebo; Test type: Other — Dose Finding; Mean Difference (Net) = -3.54, 95% CI 2-sided [-4.54 to -2.26]
Statistical Analysis 4: Comparison: LIK066 50 mg qd vs Placebo; Test type: Other — Dose Finding; Mean Difference (Net) = -3.91, 95% CI 2-sided [-5.01 to -2.77]

2. Secondary Outcome: Responder Rates According to Percentage Decrease in Body Weight From Baseline to Week 12
Description: The responder rates according to percentage decrease in body weight either ≥ 3%, ≥ 5% or ≥ 10%, from baseline at Week 12, for the overall population and each of the subgroups (Dysglycemic and Type 2 Diabetes Mellitis (T2DM)) from Baseline to Week 12 No Statistical Analysis for >=5% and >=10% was not calculated due to division by zero
Time Frame: Baseline, Week 12
Population: Full analysis set (FAS) - includes all 126 randomized participants that took at least one dose of study drug
Measure: Number; unit: Percentage of Participants
Arm/Group | LIK066 2.5mg qd | LIK066 10mg qd | LIK066 25 mg qd | LIK066 50 mg qd | Placebo
Number analyzed (Participants) | 19 | 19 | 28 | 31 | 29
Percentage of Participants
  >= 3%: number analyzed (Participants) | 19 | 18 | 28 | 30 | 28
  >= 3% | 15.8 | 55.6 | 50.0 | 56.7 | 7.1
  >= 5%: number analyzed (Participants) | 19 | 18 | 28 | 30 | 28
  >= 5% | 5.3 | 27.8 | 17.9 | 26.7 | 0.0
  >= 10%: number analyzed (Participants) | 19 | 18 | 28 | 30 | 28
  >= 10% | 0.0 | 0.0 | 0.0 | 3.3 | 0.0
  >= 3% (Dysglycemic): number analyzed (Participants) | 8 | 8 | 13 | 13 | 13
  >= 3% (Dysglycemic) | 12.5 | 75.0 | 38.5 | 46.2 | 7.7
  >= 5% (Dysglycemic): number analyzed (Participants) | 8 | 5 | 13 | 13 | 13
  >= 5% (Dysglycemic) | 0.0 | 62.5 | 23.1 | 23.1 | 0.0
  >= 10% (Dysglycemic): number analyzed (Participants) | 8 | 8 | 13 | 13 | 13
  >= 10% (Dysglycemic) | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  >= 3% (T2DM): number analyzed (Participants) | 11 | 10 | 15 | 17 | 15
  >= 3% (T2DM) | 18.2 | 40.0 | 60.0 | 64.7 | 6.7
  >= 5% (T2DM): number analyzed (Participants) | 11 | 10 | 15 | 17 | 15
  >= 5% (T2DM) | 9.1 | 0.00 | 13.3 | 29.4 | 0.00
  >= 10% (T2DM): number analyzed (Participants) | 11 | 10 | 15 | 17 | 15
  >= 10% (T2DM) | 0.00 | 0.00 | 0.00 | 5.9 | 0.00
Statistical Analysis 1: Comparison: LIK066 2.5mg qd vs Placebo; >= 3% Percent decrease in body weight; Test type: Other — Dose Finding; p = 0.390, Regression, Logistic; Odds Ratio (OR) = 2.299, 95% CI 2-sided [0.344 to 15.350]
Statistical Analysis 2: Comparison: LIK066 10mg qd vs Placebo; >= 3% Percent decrease in body weight; Test type: Other — Dose Finding; p = 0.002, Regression, Logistic; Odds Ratio (OR) = 15.780, 95% CI 2-sided [2.844 to 87.552]
Statistical Analysis 3: Comparison: LIK066 25 mg qd vs Placebo; >= 3% Percent decrease in body weight; Test type: Other — Dose Finding; p = 0.002, Regression, Logistic; Odds Ratio (OR) = 12.708, 95% CI 2-sided [2.511 to 64.320]
Statistical Analysis 4: Comparison: LIK066 50 mg qd vs Placebo; >= 3% Percent decrease in body weight; Test type: Other — Dose Finding; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 16.813, 95% CI 2-sided [3.362 to 84.085]
Statistical Analysis 5: Comparison: LIK066 2.5mg qd vs Placebo; >= 3% Percent decrease in body weight (Dysglycemic); Test type: Other — Dose Finding; p = 0.727, Regression, Logistic; Odds Ratio (OR) = 1.697, 95% CI 2-sided [0.087 to 33.006]
Statistical Analysis 6: Comparison: LIK066 10mg qd vs Placebo; >= 3% Percent decrease in body weight (Dysglycemic); Test type: Other — Dose Finding; p = 0.012, Regression, Logistic; Odds Ratio (OR) = 28.260, 95% CI 2-sided [2.066 to 386.473]
Statistical Analysis 7: Comparison: LIK066 25 mg qd vs Placebo; >= 3% Percent decrease in body weight (Dysglycemic); Test type: Other — Dose Finding; p = 0.059, Regression, Logistic; Odds Ratio (OR) = 10.333, 95% CI 2-sided [0.914 to 116.820]
Statistical Analysis 8: Comparison: LIK066 50 mg qd vs Placebo; >= 3% Percent decrease in body weight (Dysglycemic); Test type: Other — Dose Finding; p = 0.062, Regression, Logistic; Odds Ratio (OR) = 9.456, 95% CI 2-sided [0.891 to 100.292]
Statistical Analysis 9: Comparison: LIK066 2.5mg qd vs Placebo; >= 3% Percent decrease in body weight (T2DM); Test type: Other — Dose Finding; p = 0.336, Regression, Logistic; Odds Ratio (OR) = 3.590, 95% CI 2-sided [0.265 to 48.552]
Statistical Analysis 10: Comparison: LIK066 10mg qd vs Placebo; >= 3% Percent decrease in body weight (T2DM); Test type: Other — Dose Finding; p = 0.075, Regression, Logistic; Odds Ratio, log = 9.112, 95% CI 2-sided [0.799 to 103.872]
Statistical Analysis 11: Comparison: LIK066 25 mg qd vs Placebo; >= 3% Percent decrease in body weight (T2DM); Test type: Other — Dose Finding; p = 0.006, Regression, Logistic; Odds Ratio (OR) = 29.312, 95% CI 2-sided [2.665 to 322.412]
Statistical Analysis 12: Comparison: LIK066 50 mg qd vs Placebo; >= 3% Percent decrease in body weight (T2DM); Test type: Other — Dose Finding; p = 0.003, Regression, Logistic; Odds Ratio (OR) = 37.949, 95% CI 2-sided [3.477 to 414.232]

3. Secondary Outcome: Percentage Change From Baseline in Body Weight at Week 12 in Dysglycemic Participants and Participants With Type 2 Diabetes Mellitus (T2DM)
Description: The dose-response relationship for weight loss in dysglycemic participants and participants with T2DM. Percentage change from baseline in body weight at Week 12.
Time Frame: Baseline, Week 12
Population: Full analysis set (FAS) - includes all 126 randomized participants that took at least one dose of study (two subgroups Dysglycemic had total of 57 patients and T2DM had total of 69 patients) to equal 126
Measure: Number (95% Confidence Interval); unit: percentage change
Arm/Group | LIK066 2.5mg qd | LIK066 10mg qd | LIK066 25 mg qd | LIK066 50 mg qd | Placebo
Number analyzed (Participants) | 19 | 19 | 28 | 31 | 29
percentage change
  Dysglycemic: number analyzed (Participants) | 8 | 9 | 13 | 13 | 14
  Dysglycemic | -1.90 [-3.17 to -0.37] | -2.95 [-3.95 to -2.15] | -3.29 [-4.19 to -2.57] | -3.47 [-4.31 to -2.54] | 0.00 [-1.25 to 1.19]
  T2DM: number analyzed (Participants) | 11 | 10 | 15 | 18 | 15
  T2DM | -1.64 [-2.54 to -0.26] | -2.66 [-3.49 to -1.16] | -3.42 [-4.30 to -2.42] | -4.23 [-5.63 to -3.27] | 0.10 [-1.40 to 1.48]
Statistical Analysis 1: Comparison: LIK066 2.5mg qd vs Placebo; Dysglycemic; Test type: Other — Dose Finding; Median Difference (Final Values) = -1.84, 95% CI 2-sided [-3.56 to -0.19]
Statistical Analysis 2: Comparison: LIK066 10mg qd vs Placebo; Dysglycemic; Test type: Other — Dose Finding; Mean Difference (Final Values) = -2.98, 95% CI 2-sided [-4.56 to -1.46]
Statistical Analysis 3: Comparison: LIK066 25 mg qd vs Placebo; Dysglycemic; Test type: Other — Dose Finding; Mean Difference (Final Values) = -3.33, 95% CI 2-sided [-4.71 to -1.82]
Statistical Analysis 4: Comparison: LIK066 50 mg qd vs Placebo; Dysglycemic; Test type: Other — Dose Finding; Mean Difference (Final Values) = -3.51, 95% CI 2-sided [-4.93 to -1.74]
Statistical Analysis 5: Comparison: LIK066 2.5mg qd vs Placebo; T2DM; Test type: Other — Dose Finding; Mean Difference (Final Values) = -1.96, 95% CI 2-sided [-3.12 to -0.15]
Statistical Analysis 6: Comparison: LIK066 10mg qd vs Placebo; T2DM; Test type: Other — Dose Finding; Mean Difference (Final Values) = -2.88, 95% CI 2-sided [-4.37 to -0.61]
Statistical Analysis 7: Comparison: LIK066 25 mg qd vs Placebo; T2DM; Test type: Other — Dose Finding; Mean Difference (Final Values) = -3.64, 95% CI 2-sided [-5.20 to -1.52]
Statistical Analysis 8: Comparison: LIK066 50 mg qd vs Placebo; T2DM; Test type: Other — Dose Finding; Median Difference (Final Values) = -4.37, 95% CI 2-sided [-5.93 to -2.79]

4. Secondary Outcome: Change From Baseline at Week 12 on Waist Circumference at Umbilical Level
Description: Waist circumference will be measured to the nearest 0.1 cm in a standing position, at the end of a normal expiration, using a tape at the level of umbilicus. For the overall population and each of the subgroups (Dysglycemic and Type 2 Diabetes Mellitis (T2DM)) from Baseline to Week 12
Time Frame: Baseline, Week 12
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: cm
Arm/Group | LIK066 2.5mg qd | LIK066 10mg qd | LIK066 25 mg qd | LIK066 50 mg qd | Placebo
Number analyzed (Participants) | 19 | 19 | 28 | 31 | 29
cm
  Overall Study: number analyzed (Participants) | 19 | 18 | 28 | 30 | 28
  Overall Study | -2.47 [-4.003 to -0.937] | -2.63 [-4.172 to -1.082] | -2.65 [-3.907 to -1.393] | -3.11 [-4.320 to -1.895] | -1.37 [-2.636 to -0.100]
  Dysglycemic: number analyzed (Participants) | 8 | 8 | 13 | 13 | 13
  Dysglycemic | -2.78 [-5.187 to -0.368] | -4.49 [-6.856 to -2.123] | -2.08 [-3.977 to -0.177] | -2.23 [-4.123 to -0.333] | -0.41 [-2.312 to 1.483]
  T2DM: number analyzed (Participants) | 11 | 10 | 15 | 17 | 15
  T2DM | -2.22 [-4.156 to -0.283] | -1.39 [-3.418 to 0.631] | -2.90 [-4.557 to -1.244] | -3.88 [-5.416 to -2.340] | -2.19 [-3.859 to -0.520]
Statistical Analysis 1: Comparison: LIK066 2.5mg qd vs Placebo; Overall Study; Test type: Other — Dose Finding; p = 0.278, ANCOVA; Mean Difference (Final Values) = -1.10, 95% CI 2-sided [-3.104 to 0.900], Standard Error of Mean 1.011
Statistical Analysis 2: Comparison: LIK066 10mg qd vs Placebo; Overall Study; Test type: Other — Dose Finding; p = 0.216, ANCOVA; Mean Difference (Final Values) = -1.26, 95% CI 2-sided [-3.265 to 0.747], Standard Error of Mean 1.013
Statistical Analysis 3: Comparison: LIK066 25 mg qd vs Placebo; Overall Study; Test type: Other — Dose Finding; p = 0.158, ANCOVA; Mean Difference (Final Values) = -1.28, 95% CI 2-sided [-3.069 to 0.504], Standard Error of Mean 0.902
Statistical Analysis 4: Comparison: LIK066 50 mg qd vs Placebo; Overall Study; Test type: Other — Dose Finding; p = 0.053, ANCOVA; Mean Difference (Final Values) = -1.74, 95% CI 2-sided [-3.401 to 0.022], Standard Error of Mean 0.890
Statistical Analysis 5: Comparison: LIK066 2.5mg qd vs Placebo; Dysglycemic; Test type: Other — Dose Finding; p = 0.130, ANCOVA; Mean Difference (Final Values) = -2.36, 95% CI 2-sided [-5.444 to 0.717], Standard Error of Mean 1.534
Statistical Analysis 6: Comparison: LIK066 10mg qd vs Placebo; Dysglycemic; Test type: Other — Dose Finding; p = 0.011, ANCOVA; Mean Difference (Final Values) = -4.08, 95% CI 2-sided [-7.156 to -0.994], Standard Error of Mean 1.534
Statistical Analysis 7: Comparison: LIK066 25 mg qd vs Placebo; Dysglycemic; Test type: Other — Dose Finding; p = 0.215, ANCOVA; Mean Difference (Final Values) = -1.66, 95% CI 2-sided [-4.322 to 0.996], Standard Error of Mean 1.325
Statistical Analysis 8: Comparison: LIK066 50 mg qd vs Placebo; Dysglycemic; Test type: Other — Dose Finding; p = 0.184, ANCOVA; Mean Difference (Final Values) = -1.81, 95% CI 2-sided [-4.515 to 0.888], Standard Error of Mean 1.346
Statistical Analysis 9: Comparison: LIK066 2.5mg qd vs Placebo; T2DM; Test type: Other — Dose Finding; p = 0.982, ANCOVA; Mean Difference (Final Values) = -0.03, 95% CI 2-sided [-2.611 to 2.552], Standard Error of Mean 1.292
Statistical Analysis 10: Comparison: LIK066 10mg qd vs Placebo; T2DM; Test type: Other — Dose Finding; p = 0.544, ANCOVA; Mean Difference (Final Values) = 0.80, 95% CI 2-sided [-1.809 to 3.401], Standard Error of Mean 1.304
Statistical Analysis 11: Comparison: LIK066 25 mg qd vs Placebo; T2DM; Test type: Other — Dose Finding; p = 0.552, ANCOVA; Mean Difference (Final Values) = -0.71, 95% CI 2-sided [-3.084 to 1.663], Standard Error of Mean 1.188
Statistical Analysis 12: Comparison: LIK066 50 mg qd vs Placebo; T2DM; Test type: Other — Dose Finding; p = 0.143, ANCOVA; Mean Difference (Final Values) = -1.69, 95% CI 2-sided [-3.964 to 0.588], Standard Error of Mean 1.139

5. Secondary Outcome: Percentage Change From Baseline at Week 12 on Hemoglobin A1c (HbA1c)
Description: HbA1c will be measured from a blood sample obtained and analyzed at a central laboratory. For the overall population and each of the subgroups (Dysglycemic and Type 2 Diabetes Mellitis (T2DM)) from Baseline to Week 12
Time Frame: Baseline, Week 12
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: Percentage
Arm/Group | LIK066 2.5mg qd | LIK066 10mg qd | LIK066 25 mg qd | LIK066 50 mg qd | Placebo
Number analyzed (Participants) | 19 | 19 | 28 | 31 | 29
Percentage
  Overall Study: number analyzed (Participants) | 19 | 18 | 28 | 30 | 28
  Overall Study | -0.285 [-0.415 to -0.155] | -0.355 [-0.488 to -0.223] | -0.366 [-0.473 to -0.259] | -0.418 [-0.521 to -0.314] | -0.079 [-0.187 to 0.028]
  Dysglycemic: number analyzed (Participants) | 8 | 8 | 13 | 13 | 13
  Dysglycemic | -0.139 [-0.261 to -0.016] | -0.184 [-0.306 to -0.062] | -0.196 [-0.292 to -0.101] | -0.163 [-0.259 to -0.067] | -0.050 [-0.146 to 0.046]
  T2DM: number analyzed (Participants) | 11 | 10 | 15 | 17 | 15
  T2DM | -0.405 [-0.616 to -0.195] | -0.491 [-0.708 to -0.275] | -0.502 [-0.679 to -0.325] | -0.618 [-0.784 to -0.452] | -0.093 [-0.271 to 0.086]
Statistical Analysis 1: Comparison: LIK066 2.5mg qd vs Placebo; Overall Study; Test type: Other — Dose Finding; p = 0.018, ANCOVA; Mean Difference (Final Values) = -0.206, 95% CI 2-sided [-0.376 to -0.035], Standard Error of Mean 0.0860
Statistical Analysis 2: Comparison: LIK066 10mg qd vs Placebo; Overall Study; Test type: Other — Dose Finding; p = 0.002, ANCOVA; Mean Difference (Final Values) = -0.276, 95% CI 2-sided [-0.447 to -0.105], Standard Error of Mean 0.0863
Statistical Analysis 3: Comparison: LIK066 25 mg qd vs Placebo; Overall Study; Test type: Other — Dose Finding; p < 0.001, ANCOVA; Mean Difference (Final Values) = -0.287, 95% CI 2-sided [-0.437 to -0.136], Standard Error of Mean 0.0760
Statistical Analysis 4: Comparison: LIK066 50 mg qd vs Placebo; Overall Study; Test type: Other — Dose Finding; p < 0.001, ANCOVA; Mean Difference (Final Values) = -0.338, 95% CI 2-sided [-0.486 to -0.190], Standard Error of Mean 0.0747
Statistical Analysis 5: Comparison: LIK066 2.5mg qd vs Placebo; Dysglycemic; Test type: Other — Dose Finding; p = 0.258, ANCOVA; Mean Difference (Final Values) = -0.089, 95% CI 2-sided [-0.245 to 0.067], Standard Error of Mean 0.0775
Statistical Analysis 6: Comparison: LIK066 10mg qd vs Placebo; Dysglycemic; Test type: Other — Dose Finding; p = 0.088, ANCOVA; Mean Difference (Final Values) = -0.134, 95% CI 2-sided [-0.290 to 0.021], Standard Error of Mean 0.0774
Statistical Analysis 7: Comparison: LIK066 25 mg qd vs Placebo; Dysglycemic; Test type: Other — Dose Finding; p = 0.035, ANCOVA; Mean Difference (Final Values) = -0.146, 95% CI 2-sided [-0.282 to -0.011], Standard Error of Mean 0.0673
Statistical Analysis 8: Comparison: LIK066 50 mg qd vs Placebo; Dysglycemic; Test type: Other — Dose Finding; p = 0.100, ANCOVA; Mean Difference (Final Values) = -0.113, 95% CI 2-sided [-0.248 to 0.022], Standard Error of Mean 0.0673
Statistical Analysis 9: Comparison: LIK066 2.5mg qd vs Placebo; T2DM; Test type: Other — Dose Finding; p = 0.029, ANCOVA; Mean Difference (Final Values) = -0.313, 95% CI 2-sided [-0.592 to -0.033], Standard Error of Mean 0.1399
Statistical Analysis 10: Comparison: LIK066 10mg qd vs Placebo; T2DM; Test type: Other — Dose Finding; p = 0.006, ANCOVA; Mean Difference (Final Values) = -0.399, 95% CI 2-sided [-0.681 to -0.117], Standard Error of Mean 0.1411
Statistical Analysis 11: Comparison: LIK066 25 mg qd vs Placebo; T2DM; Test type: Other — Dose Finding; p = 0.002, ANCOVA; Mean Difference (Final Values) = -0.409, 95% CI 2-sided [-0.660 to -0.159], Standard Error of Mean 0.1253
Statistical Analysis 12: Comparison: LIK066 50 mg qd vs Placebo; T2DM; Test type: Other — Dose Finding; p < 0.001, ANCOVA; Mean Difference (Final Values) = -0.526, 95% CI 2-sided [-0.769 to -0.282], Standard Error of Mean 0.1217

6. Secondary Outcome: Change From Baseline at Week 12 on Fasting Plasma Glucose (FPG)
Description: FPG will be measured from a blood sample obtained after an overnight fast (at least 8h after last evening food intake) at a central laboratory. For the overall population and each of the subgroups (Dysglycemic and Type 2 Diabetes Mellitis (T2DM)) from Baseline to Week 12
Time Frame: Baseline, Week 12
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | LIK066 2.5mg qd | LIK066 10mg qd | LIK066 25 mg qd | LIK066 50 mg qd | Placebo
Number analyzed (Participants) | 19 | 19 | 28 | 31 | 29
mmol/L
  Overall Study: number analyzed (Participants) | 19 | 18 | 28 | 30 | 28
  Overall Study | -0.334 [-0.652 to -0.016] | -0.665 [-0.990 to -0.340] | -0.747 [-1.007 to -0.486] | -0.986 [-1.238 to -0.733] | -0.160 [-0.423 to 0.103]
  Dysglycemic: number analyzed (Participants) | 8 | 8 | 13 | 13 | 13
  Dysglycemic | 0.002 [-0.322 to 0.326] | -0.126 [-0.453 to 0.200] | -0.262 [-0.515 to -0.008] | -0.472 [-0.728 to -0.217] | -0.217 [-0.471 to 0.038]
  T2DM: number analyzed (Participants) | 11 | 10 | 15 | 17 | 15
  T2DM | -0.606 [-1.095 to -0.118] | -1.111 [-1.619 to -0.604] | -1.145 [-1.559 to -0.730] | -1.377 [-1.766 to -0.988] | -0.079 [-0.497 to 0.339]
Statistical Analysis 1: Comparison: LIK066 2.5mg qd vs Placebo; Overall Study; Test type: Other — Dose Finding; p = 0.408, ANCOVA; Mean Difference (Final Values) = -0.174, 95% CI 2-sided [-0.589 to 0.241], Standard Error of Mean 0.2094
Statistical Analysis 2: Comparison: LIK066 10mg qd vs Placebo; Overall Study; Test type: Other — Dose Finding; p = 0.018, ANCOVA; Mean Difference (Final Values) = -0.505, 95% CI 2-sided [-0.924 to -0.087], Standard Error of Mean 0.2115
Statistical Analysis 3: Comparison: LIK066 25 mg qd vs Placebo; Overall Study; Test type: Other — Dose Finding; p = 0.002, ANCOVA; Mean Difference (Final Values) = -0.587, 95% CI 2-sided [-0.956 to -0.217], Standard Error of Mean 0.1866
Statistical Analysis 4: Comparison: LIK066 50 mg qd vs Placebo; Overall Study; Test type: Other — Dose Finding; p < 0.001, ANCOVA; Mean Difference (Final Values) = -0.826, 95% CI 2-sided [-1.188 to -0.463], Standard Error of Mean 0.1831
Statistical Analysis 5: Comparison: LIK066 2.5mg qd vs Placebo; Dysglycemic; Test type: Other — Dose Finding; p = 0.293, ANCOVA; Mean Difference (Final Values) = 0.218, 95% CI 2-sided [-0.194 to 0.631], Standard Error of Mean 0.2054
Statistical Analysis 6: Comparison: LIK066 10mg qd vs Placebo; Dysglycemic; Test type: Other — Dose Finding; p = 0.665, ANCOVA; Mean Difference (Final Values) = 0.090, 95% CI 2-sided [-0.325 to 0.506], Standard Error of Mean 0.2068
Statistical Analysis 7: Comparison: LIK066 25 mg qd vs Placebo; Dysglycemic; Test type: Other — Dose Finding; p = 0.803, ANCOVA; Mean Difference (Final Values) = -0.045, 95% CI 2-sided [-0.405 to 0.315], Standard Error of Mean 0.1791
Statistical Analysis 8: Comparison: LIK066 50 mg qd vs Placebo; Dysglycemic; Test type: Other — Dose Finding; p = 0.159, ANCOVA; Mean Difference (Final Values) = -0.256, 95% CI 2-sided [-0.615 to 0.103], Standard Error of Mean 0.1787
Statistical Analysis 9: Comparison: LIK066 2.5mg qd vs Placebo; T2DM; Test type: Other — Dose Finding; p = 0.110, ANCOVA; Mean Difference (Final Values) = -0.527, 95% CI 2-sided [-1.176 to 0.122], Standard Error of Mean 0.3249
Statistical Analysis 10: Comparison: LIK066 10mg qd vs Placebo; T2DM; Test type: Other — Dose Finding; p = 0.003, ANCOVA; Mean Difference (Final Values) = -1.032, 95% CI 2-sided [-1.691 to -0.373], Standard Error of Mean 0.3296
Statistical Analysis 11: Comparison: LIK066 25 mg qd vs Placebo; T2DM; Test type: Other — Dose Finding; p < 0.001, ANCOVA; Mean Difference (Final Values) = -1.065, 95% CI 2-sided [-1.654 to -0.476], Standard Error of Mean 0.2946
Statistical Analysis 12: Comparison: LIK066 50 mg qd vs Placebo; T2DM; Test type: Other — Dose Finding; p < 0.001, ANCOVA; Mean Difference (Final Values) = -1.298, 95% CI 2-sided [-1.869 to -0.728], Standard Error of Mean 0.2855

7. Secondary Outcome: Change From Baseline at Week 12 on Systolic Blood Pressure (SBP)
Description: After the subject has been sitting for 5 minutes with the back supported and both feet placed on the floor, SBP will be measured three times using the automatic BP monitor and an appropriate size cuff. For the overall population and each of the subgroups (Dysglycemic and Type 2 Diabetes Mellitis (T2DM)) from Baseline to Week 12
Time Frame: Baseline, Week 12
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | LIK066 2.5mg qd | LIK066 10mg qd | LIK066 25 mg qd | LIK066 50 mg qd | Placebo
Number analyzed (Participants) | 19 | 19 | 28 | 31 | 29
mmHg
  Overall Study: number analyzed (Participants) | 19 | 18 | 28 | 30 | 28
  Overall Study | -4.90 [-9.049 to -0.746] | -5.12 [-9.403 to -0.834] | -6.36 [-9.781 to -2.935] | -6.94 [-10.233 to -3.655] | -5.36 [-8.758 to -1.961]
  Dysglycemic: number analyzed (Participants) | 8 | 8 | 13 | 13 | 13
  Dysglycemic | -5.79 [-12.457 to 0.883] | -7.10 [-13.825 to -0.369] | -3.58 [-8.811 to 1.657] | -4.17 [-9.399 to 1.051] | -7.09 [-12.294 to -1.891]
  T2DM: number analyzed (Participants) | 11 | 10 | 15 | 17 | 15
  T2DM | -4.16 [-9.414 to 1.091] | -2.96 [-8.500 to 2.588] | -8.63 [-13.143 to -4.120] | -9.00 [-13.182 to -4.810] | -3.77 [-8.255 to 0.724]
Statistical Analysis 1: Comparison: LIK066 2.5mg qd vs Placebo; Overall Study; Test type: Other — Dose Finding; p = 0.865, ANCOVA; Mean Difference (Final Values) = 0.46, 95% CI 2-sided [-4.898 to 5.822], Standard Error of Mean 2.707
Statistical Analysis 2: Comparison: LIK066 10mg qd vs Placebo; Overall Study; Test type: Other — Dose Finding; p = 0.931, ANCOVA; Mean Difference (Final Values) = 0.24, 95% CI 2-sided [-5.235 to 5.716], Standard Error of Mean 2.765
Statistical Analysis 3: Comparison: LIK066 25 mg qd vs Placebo; Overall Study; Test type: Other — Dose Finding; p = 0.682, ANCOVA; Mean Difference (Final Values) = -1.00, 95% CI 2-sided [-5.817 to 3.820], Standard Error of Mean 2.433
Statistical Analysis 4: Comparison: LIK066 50 mg qd vs Placebo; Overall Study; Test type: Other — Dose Finding; p = 0.508, ANCOVA; Mean Difference (Final Values) = -1.58, 95% CI 2-sided [-6.312 to 3.142], Standard Error of Mean 2.387
Statistical Analysis 5: Comparison: LIK066 2.5mg qd vs Placebo; Dysglycemic; Test type: Other — Dose Finding; p = 0.757, ANCOVA; Mean Difference (Final Values) = 1.31, 95% CI 2-sided [-7.138 to 9.749], Standard Error of Mean 4.206
Statistical Analysis 6: Comparison: LIK066 10mg qd vs Placebo; Dysglycemic; Test type: Other — Dose Finding; p = 0.999, ANCOVA; Mean Difference (Final Values) = 0.00, 95% CI 2-sided [-8.571 to 8.563], Standard Error of Mean 4.267
Statistical Analysis 7: Comparison: LIK066 25 mg qd vs Placebo; Dysglycemic; Test type: Other — Dose Finding; p = 0.342, ANCOVA; Mean Difference (Final Values) = 3.52, 95% CI 2-sided [-3.848 to 10.880], Standard Error of Mean 3.668
Statistical Analysis 8: Comparison: LIK066 50 mg qd vs Placebo; Dysglycemic; Test type: Other — Dose Finding; p = 0.430, ANCOVA; Mean Difference (Final Values) = 2.92, 95% CI 2-sided [-4.454 to 10.292], Standard Error of Mean 3.673
Statistical Analysis 9: Comparison: LIK066 2.5mg qd vs Placebo; T2DM; Test type: Other — Dose Finding; p = 0.909, ANCOVA; Mean Difference (Final Values) = -0.40, 95% CI 2-sided [-7.312 to 6.520], Standard Error of Mean 3.461
Statistical Analysis 10: Comparison: LIK066 10mg qd vs Placebo; T2DM; Test type: Other — Dose Finding; p = 0.821, ANCOVA; Mean Difference (Final Values) = 0.81, 95% CI 2-sided [-6.311 to 7.930], Standard Error of Mean 3.563
Statistical Analysis 11: Comparison: LIK066 25 mg qd vs Placebo; T2DM; Test type: Other — Dose Finding; p = 0.132, ANCOVA; Mean Difference (Final Values) = -4.87, 95% CI 2-sided [-11.240 to 1.508], Standard Error of Mean 3.190
Statistical Analysis 12: Comparison: LIK066 50 mg qd vs Placebo; T2DM; Test type: Other — Dose Finding; p = 0.093, ANCOVA; Mean Difference (Final Values) = -5.23, 95% CI 2-sided [-11.367 to 0.905], Standard Error of Mean 3.070

8. Secondary Outcome: Change From Baseline at Week 12 on Diastolic Blood Pressure (DBP)
Description: After the subject has been sitting for 5 minutes with the back supported and both feet placed on the floor, DBP will be measured three times using the automatic BP monitor and an appropriate size cuff. For the overall population and each of the subgroups (Dysglycemic and Type 2 Diabetes Mellitis (T2DM)) from Baseline to Week 12
Time Frame: Baseline, Week 12
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | LIK066 2.5mg qd | LIK066 10mg qd | LIK066 25 mg qd | LIK066 50 mg qd | Placebo
Number analyzed (Participants) | 19 | 19 | 28 | 31 | 29
mmHg
  Overall Study: number analyzed (Participants) | 19 | 18 | 28 | 30 | 28
  Overall Study | -3.72 [-6.803 to -0.627] | -3.54 [-6.700 to -0.377] | -4.36 [-6.892 to -1.818] | -5.23 [-7.677 to -2.788] | -3.12 [-5.647 to -0.597]
  Dysglycemic: number analyzed (Participants) | 8 | 8 | 13 | 13 | 13
  Dysglycemic | -3.32 [-8.404 to 1.769] | -4.40 [-9.490 to 0.699] | -2.46 [-6.441 to 1.513] | -4.25 [-8.230 to -0.279] | -4.31 [-8.257 to -0.357]
  T2DM: number analyzed (Participants) | 11 | 10 | 15 | 17 | 15
  T2DM | -4.00 [-7.943 to -0.059] | -2.45 [-6.584 to 1.687] | -5.98 [-9.352 to -2.607] | -5.92 [-9.066 to -2.776] | -1.93 [-5.303 to 1.448]
Statistical Analysis 1: Comparison: LIK066 2.5mg qd vs Placebo; Overall Study; Test type: Other — Dose Finding; p = 0.769, ANCOVA; Mean Difference (Final Values) = -0.59, 95% CI 2-sided [-4.579 to 3.393], Standard Error of Mean 2.013
Statistical Analysis 2: Comparison: LIK066 10mg qd vs Placebo; Overall Study; Test type: Other — Dose Finding; p = 0.839, ANCOVA; Mean Difference (Final Values) = -0.42, 95% CI 2-sided [-4.462 to 3.630], Standard Error of Mean 2.043
Statistical Analysis 3: Comparison: LIK066 25 mg qd vs Placebo; Overall Study; Test type: Other — Dose Finding; p = 0.496, ANCOVA; Mean Difference (Final Values) = -1.23, 95% CI 2-sided [-4.811 to 2.345], Standard Error of Mean 1.807
Statistical Analysis 4: Comparison: LIK066 50 mg qd vs Placebo; Overall Study; Test type: Other — Dose Finding; p = 0.237, ANCOVA; Mean Difference (Final Values) = -2.11, 95% CI 2-sided [-5.622 to 1.402], Standard Error of Mean 1.774
Statistical Analysis 5: Comparison: LIK066 2.5mg qd vs Placebo; Dysglycemic; Test type: Other — Dose Finding; p = 0.758, ANCOVA; Mean Difference (Final Values) = 0.99, 95% CI 2-sided [-5.435 to 7.415], Standard Error of Mean 3.200
Statistical Analysis 6: Comparison: LIK066 10mg qd vs Placebo; Dysglycemic; Test type: Other — Dose Finding; p = 0.978, ANCOVA; Mean Difference (Final Values) = -0.09, 95% CI 2-sided [-6.574 to 6.397], Standard Error of Mean 3.230
Statistical Analysis 7: Comparison: LIK066 25 mg qd vs Placebo; Dysglycemic; Test type: Other — Dose Finding; p = 0.512, ANCOVA; Mean Difference (Final Values) = 1.84, 95% CI 2-sided [-3.758 to 7.444], Standard Error of Mean 2.790
Statistical Analysis 8: Comparison: LIK066 50 mg qd vs Placebo; Dysglycemic; Test type: Other — Dose Finding; p = 0.985, ANCOVA; Mean Difference (Final Values) = 0.05, 95% CI 2-sided [-5.552 to 5.657], Standard Error of Mean 2.792
Statistical Analysis 9: Comparison: LIK066 2.5mg qd vs Placebo; T2DM; Test type: Other — Dose Finding; p = 0.428, ANCOVA; Mean Difference (Final Values) = -2.07, 95% CI 2-sided [-7.268 to 3.121], Standard Error of Mean 2.599
Statistical Analysis 10: Comparison: LIK066 10mg qd vs Placebo; T2DM; Test type: Other — Dose Finding; p = 0.846, ANCOVA; Mean Difference (Final Values) = -0.52, 95% CI 2-sided [-5.853 to 4.812], Standard Error of Mean 2.669
Statistical Analysis 11: Comparison: LIK066 25 mg qd vs Placebo; T2DM; Test type: Other — Dose Finding; p = 0.095, ANCOVA; Mean Difference (Final Values) = -4.05, 95% CI 2-sided [-8.825 to 0.721], Standard Error of Mean 2.388
Statistical Analysis 12: Comparison: LIK066 50 mg qd vs Placebo; T2DM; Test type: Other — Dose Finding; p = 0.089, ANCOVA; Mean Difference (Final Values) = -3.99, 95% CI 2-sided [-8.610 to 0.623], Standard Error of Mean 2.310

9. Secondary Outcome: Percentage Change From Baseline at Week 12 on Fasting Lipid Profile - Triglycerides (TG)
Description: Fasting lipid profile (Triglycerides (TG)), will be measured on blood samples obtained after an overnight fast and analyzed at a central laboratory For the overall population and each of the subgroups (Dysglycemic and Type 2 Diabetes Mellitis (T2DM)) from Baseline to Week 12
Time Frame: Baseline, Week 12
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: Percentage
Arm/Group | LIK066 2.5mg qd | LIK066 10mg qd | LIK066 25 mg qd | LIK066 50 mg qd | Placebo
Number analyzed (Participants) | 19 | 19 | 28 | 31 | 29
Percentage
  Overall Study: number analyzed (Participants) | 19 | 18 | 28 | 30 | 28
  Overall Study | 1.840 [-30.956 to 34.636] | 11.057 [-22.372 to 44.487] | 43.928 [17.118 to 70.737] | 5.307 [-20.648 to 31.261] | 17.401 [-9.474 to 44.275]
  Dysglycemic: number analyzed (Participants) | 8 | 8 | 13 | 13 | 13
  Dysglycemic | -1.153 [-62.637 to 60.331] | -1.986 [-64.104 to 60.132] | 52.284 [3.839 to 100.729] | 14.061 [-34.625 to 62.746] | 20.962 [-27.416 to 69.340]
  T2DM: number analyzed (Participants) | 11 | 10 | 15 | 17 | 15
  T2DM | 1.016 [-36.069 to 38.100] | 23.108 [-14.937 to 61.153] | 34.747 [3.600 to 65.893] | -0.057 [-29.478 to 29.363] | 13.806 [-17.085 to 44.697]
Statistical Analysis 1: Comparison: LIK066 2.5mg qd vs Placebo; Overall Study; Test type: Other — Dose Finding; p = 0.470, ANCOVA; Mean Difference (Final Values) = -15.561, 95% CI 2-sided [-58.106 to 26.985], Standard Error of Mean 21.4808
Statistical Analysis 2: Comparison: LIK066 10mg qd vs Placebo; Overall Study; Test type: Other — Dose Finding; p = 0.770, ANCOVA; Mean Difference (Final Values) = -6.343, 95% CI 2-sided [-49.187 to 36.501], Standard Error of Mean 21.6316
Statistical Analysis 3: Comparison: LIK066 25 mg qd vs Placebo; Overall Study; Test type: Other — Dose Finding; p = 0.169, ANCOVA; Mean Difference (Final Values) = 26.527, 95% CI 2-sided [-11.462 to 64.516], Standard Error of Mean 19.1803
Statistical Analysis 4: Comparison: LIK066 50 mg qd vs Placebo; Overall Study; Test type: Other — Dose Finding; p = 0.521, ANCOVA; Mean Difference (Final Values) = -12.094, 95% CI 2-sided [-49.345 to 25.157], Standard Error of Mean 18.8076
Statistical Analysis 5: Comparison: LIK066 2.5mg qd vs Placebo; Dysglycemic; Test type: Other — Dose Finding; p = 0.571, ANCOVA; Mean Difference (Final Values) = -22.115, 95% CI 2-sided [-100.058 to 55.828], Standard Error of Mean 38.7858
Statistical Analysis 6: Comparison: LIK066 10mg qd vs Placebo; Dysglycemic; Test type: Other — Dose Finding; p = 0.564, ANCOVA; Mean Difference (Final Values) = -22.948, 95% CI 2-sided [-102.325 to 56.429], Standard Error of Mean 39.4994
Statistical Analysis 7: Comparison: LIK066 25 mg qd vs Placebo; Dysglycemic; Test type: Other — Dose Finding; p = 0.359, ANCOVA; Mean Difference (Final Values) = 31.322, 95% CI 2-sided [-36.712 to 99.356], Standard Error of Mean 33.8550
Statistical Analysis 8: Comparison: LIK066 50 mg qd vs Placebo; Dysglycemic; Test type: Other — Dose Finding; p = 0.842, ANCOVA; Mean Difference (Final Values) = -6.901, 95% CI 2-sided [-76.093 to 62.290], Standard Error of Mean 34.4309
Statistical Analysis 9: Comparison: LIK066 2.5mg qd vs Placebo; T2DM; Test type: Other — Dose Finding; p = 0.601, ANCOVA; Mean Difference (Final Values) = -12.790, 95% CI 2-sided [-61.417 to 35.836], Standard Error of Mean 24.3259
Statistical Analysis 10: Comparison: LIK066 10mg qd vs Placebo; T2DM; Test type: Other — Dose Finding; p = 0.705, ANCOVA; Mean Difference (Final Values) = 9.302, 95% CI 2-sided [-39.517 to 58.121], Standard Error of Mean 24.4220
Statistical Analysis 11: Comparison: LIK066 25 mg qd vs Placebo; T2DM; Test type: Other — Dose Finding; p = 0.346, ANCOVA; Mean Difference (Final Values) = 20.940, 95% CI 2-sided [-23.126 to 65.007], Standard Error of Mean 22.0444
Statistical Analysis 12: Comparison: LIK066 50 mg qd vs Placebo; T2DM; Test type: Other — Dose Finding; p = 0.516, ANCOVA; Mean Difference (Final Values) = -13.863, 95% CI 2-sided [-56.283 to 28.556], Standard Error of Mean 21.2205

10. Secondary Outcome: Percentage Change From Baseline at Week 12 on Fasting Lipid Profile - Total Cholesterol
Description: Fasting lipid profile (total cholesterol), will be measured on blood samples obtained after an overnight fast and analyzed at a central laboratory For the overall population and each of the subgroups (Dysglycemic and Type 2 Diabetes Mellitis (T2DM)) from Baseline to Week 12
Time Frame: Baseline, Week 12
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: Percentage
Arm/Group | LIK066 2.5mg qd | LIK066 10mg qd | LIK066 25 mg qd | LIK066 50 mg qd | Placebo
Number analyzed (Participants) | 19 | 19 | 28 | 31 | 29
Percentage
  Overall Study: number analyzed (Participants) | 19 | 18 | 28 | 30 | 28
  Overall Study | -1.290 [-6.809 to 4.229] | -2.983 [-8.711 to 2.745] | 0.884 [-3.663 to 5.430] | 0.302 [-4.096 to 4.700] | -2.244 [-6.800 to 2.312]
  Dysglycemic: number analyzed (Participants) | 8 | 8 | 13 | 13 | 13
  Dysglycemic | -3.055 [-12.284 to 6.173] | -6.017 [-15.916 to 3.882] | 4.273 [-3.085 to 11.630] | -1.734 [-9.000 to 5.532] | -3.559 [-10.940 to 3.822]
  T2DM: number analyzed (Participants) | 11 | 10 | 15 | 17 | 15
  T2DM | 0.158 [-6.814 to 7.129] | -1.367 [-8.670 to 5.937] | -1.646 [-7.772 to 4.481] | 1.817 [-3.857 to 7.491] | -0.671 [-6.635 to 5.294]
Statistical Analysis 1: Comparison: LIK066 2.5mg qd vs Placebo; Overall Study; Test type: Other — Dose Finding; p = 0.792, ANCOVA; Mean Difference (Final Values) = 0.955, 95% CI 2-sided [-6.185 to 8.095], Standard Error of Mean 3.6050
Statistical Analysis 2: Comparison: LIK066 10mg qd vs Placebo; Overall Study; Test type: Other — Dose Finding; p = 0.843, ANCOVA; Mean Difference (Final Values) = -0.739, 95% CI 2-sided [-8.100 to 6.623], Standard Error of Mean 3.7167
Statistical Analysis 3: Comparison: LIK066 25 mg qd vs Placebo; Overall Study; Test type: Other — Dose Finding; p = 0.339, ANCOVA; Mean Difference (Final Values) = 3.128, 95% CI 2-sided [-3.322 to 9.578], Standard Error of Mean 3.2564
Statistical Analysis 4: Comparison: LIK066 50 mg qd vs Placebo; Overall Study; Test type: Other — Dose Finding; p = 0.426, ANCOVA; Mean Difference (Final Values) = 2.546, 95% CI 2-sided [-3.764 to 8.856], Standard Error of Mean 3.1859
Statistical Analysis 5: Comparison: LIK066 2.5mg qd vs Placebo; Dysglycemic; Test type: Other — Dose Finding; p = 0.932, ANCOVA; Mean Difference (Final Values) = 0.504, 95% CI 2-sided [-11.299 to 12.307], Standard Error of Mean 5.8734
Statistical Analysis 6: Comparison: LIK066 10mg qd vs Placebo; Dysglycemic; Test type: Other — Dose Finding; p = 0.700, ANCOVA; Mean Difference (Final Values) = -2.458, 95% CI 2-sided [-15.217 to 10.302], Standard Error of Mean 6.3493
Statistical Analysis 7: Comparison: LIK066 25 mg qd vs Placebo; Dysglycemic; Test type: Other — Dose Finding; p = 0.131, ANCOVA; Mean Difference (Final Values) = 7.832, 95% CI 2-sided [-2.406 to 18.070], Standard Error of Mean 5.0946
Statistical Analysis 8: Comparison: LIK066 50 mg qd vs Placebo; Dysglycemic; Test type: Other — Dose Finding; p = 0.727, ANCOVA; Mean Difference (Final Values) = 1.825, 95% CI 2-sided [-8.619 to 12.269], Standard Error of Mean 5.1970
Statistical Analysis 9: Comparison: LIK066 2.5mg qd vs Placebo; T2DM; Test type: Other — Dose Finding; p = 0.857, ANCOVA; Mean Difference (Final Values) = 0.828, 95% CI 2-sided [-8.342 to 9.999], Standard Error of Mean 4.5876
Statistical Analysis 10: Comparison: LIK066 10mg qd vs Placebo; T2DM; Test type: Other — Dose Finding; p = 0.883, ANCOVA; Mean Difference (Final Values) = -0.696, 95% CI 2-sided [-10.126 to 8.734], Standard Error of Mean 4.7173
Statistical Analysis 11: Comparison: LIK066 25 mg qd vs Placebo; T2DM; Test type: Other — Dose Finding; p = 0.821, ANCOVA; Mean Difference (Final Values) = -0.975, 95% CI 2-sided [-9.547 to 7.597], Standard Error of Mean 4.2883
Statistical Analysis 12: Comparison: LIK066 50 mg qd vs Placebo; T2DM; Test type: Other — Dose Finding; p = 0.547, ANCOVA; Mean Difference (Final Values) = 2.488, 95% CI 2-sided [-5.730 to 10.706], Standard Error of Mean 4.1111

11. Secondary Outcome: Percentage Change From Baseline at Week 12 on Fasting Lipid Profile - High Density Lipoprotein (HDL)
Description: Fasting lipid profile (HDL), will be measured on blood samples obtained after an overnight fast and analyzed at a central laboratory For the overall population and each of the subgroups (Dysglycemic and Type 2 Diabetes Mellitis (T2DM)) from Baseline to Week 12
Time Frame: Baseline, Week 12
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: Percentage
Arm/Group | LIK066 2.5mg qd | LIK066 10mg qd | LIK066 25 mg qd | LIK066 50 mg qd | Placebo
Number analyzed (Participants) | 19 | 19 | 28 | 31 | 29
Percentage
  Overall Study: number analyzed (Participants) | 19 | 18 | 28 | 30 | 28
  Overall Study | 1.499 [-3.683 to 6.682] | -2.461 [-7.790 to 2.868] | -5.253 [-9.514 to -0.993] | 0.112 [-4.014 to 4.237] | -3.454 [-7.739 to 0.830]
  Dysglycemic: number analyzed (Participants) | 8 | 8 | 13 | 13 | 13
  Dysglycemic | -0.519 [-9.144 to 8.107] | 0.329 [-8.368 to 9.027] | -3.279 [-10.056 to 3.498] | -0.147 [-6.917 to 6.622] | -4.329 [-11.096 to 2.437]
  T2DM: number analyzed (Participants) | 11 | 10 | 15 | 17 | 15
  T2DM | 2.886 [-3.774 to 9.545] | -4.696 [-11.654 to 2.261] | -6.993 [-12.672 to -1.315] | 0.235 [-5.133 to 5.604] | -2.677 [-8.484 to 3.130]
Statistical Analysis 1: Comparison: LIK066 2.5mg qd vs Placebo; Overall Study; Test type: Other — Dose Finding; p = 0.148, ANCOVA; Mean Difference (Final Values) = 4.954, 95% CI 2-sided [-1.781 to 11.689], Standard Error of Mean 3.4006
Statistical Analysis 2: Comparison: LIK066 10mg qd vs Placebo; Overall Study; Test type: Other — Dose Finding; p = 0.775, ANCOVA; Mean Difference (Final Values) = 0.993, 95% CI 2-sided [-5.869 to 7.855], Standard Error of Mean 3.4645
Statistical Analysis 3: Comparison: LIK066 25 mg qd vs Placebo; Overall Study; Test type: Other — Dose Finding; p = 0.556, ANCOVA; Mean Difference (Final Values) = -1.799, 95% CI 2-sided [-7.826 to 4.229], Standard Error of Mean 3.0432
Statistical Analysis 4: Comparison: LIK066 50 mg qd vs Placebo; Overall Study; Test type: Other — Dose Finding; p = 0.238, ANCOVA; Mean Difference (Final Values) = 3.566, 95% CI 2-sided [-2.391 to 9.524], Standard Error of Mean 3.0079
Statistical Analysis 5: Comparison: LIK066 2.5mg qd vs Placebo; Dysglycemic; Test type: Other — Dose Finding; p = 0.488, ANCOVA; Mean Difference (Final Values) = 3.811, 95% CI 2-sided [-7.152 to 14.774], Standard Error of Mean 5.4552
Statistical Analysis 6: Comparison: LIK066 10mg qd vs Placebo; Dysglycemic; Test type: Other — Dose Finding; p = 0.400, ANCOVA; Mean Difference (Final Values) = 4.659, 95% CI 2-sided [-6.363 to 15.680], Standard Error of Mean 5.4845
Statistical Analysis 7: Comparison: LIK066 25 mg qd vs Placebo; Dysglycemic; Test type: Other — Dose Finding; p = 0.826, ANCOVA; Mean Difference (Final Values) = 1.050, 95% CI 2-sided [-8.525 to 10.626], Standard Error of Mean 4.7651
Statistical Analysis 8: Comparison: LIK066 50 mg qd vs Placebo; Dysglycemic; Test type: Other — Dose Finding; p = 0.384, ANCOVA; Mean Difference (Final Values) = 4.182, 95% CI 2-sided [-5.389 to 13.753], Standard Error of Mean 4.7627
Statistical Analysis 9: Comparison: LIK066 2.5mg qd vs Placebo; T2DM; Test type: Other — Dose Finding; p = 0.217, ANCOVA; Mean Difference (Final Values) = 5.563, 95% CI 2-sided [-3.360 to 14.486], Standard Error of Mean 4.4636
Statistical Analysis 10: Comparison: LIK066 10mg qd vs Placebo; T2DM; Test type: Other — Dose Finding; p = 0.659, ANCOVA; Mean Difference (Final Values) = -2.019, 95% CI 2-sided [-11.112 to 7.074], Standard Error of Mean 4.5491
Statistical Analysis 11: Comparison: LIK066 25 mg qd vs Placebo; T2DM; Test type: Other — Dose Finding; p = 0.291, ANCOVA; Mean Difference (Final Values) = -4.316, 95% CI 2-sided [-12.423 to 3.791], Standard Error of Mean 4.0556
Statistical Analysis 12: Comparison: LIK066 50 mg qd vs Placebo; T2DM; Test type: Other — Dose Finding; p = 0.470, ANCOVA; Mean Difference (Final Values) = 2.913, 95% CI 2-sided [-5.090 to 10.916], Standard Error of Mean 4.0035

12. Secondary Outcome: Percentage Change From Baseline at Week 12 on Fasting Lipid Profile - Low Density Lipoprotein (LDL)
Description: Fasting lipid profile (LDL), will be measured on blood samples obtained after an overnight fast and analyzed at a central laboratory For the overall population and each of the subgroups (Dysglycemic and Type 2 Diabetes Mellitis (T2DM)) from Baseline to Week 12
Time Frame: Baseline, Week 12
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: Percentage
Arm/Group | LIK066 2.5mg qd | LIK066 10mg qd | LIK066 25 mg qd | LIK066 50 mg qd | Placebo
Number analyzed (Participants) | 19 | 19 | 28 | 31 | 29
Percentage
  Overall Study: number analyzed (Participants) | 19 | 18 | 28 | 30 | 28
  Overall Study | 0.757 [-7.220 to 8.734] | -2.363 [-10.702 to 5.975] | 0.037 [-6.524 to 6.598] | 4.726 [-1.616 to 11.068] | -0.552 [-7.154 to 6.051]
  Dysglycemic: number analyzed (Participants) | 8 | 8 | 13 | 13 | 13
  Dysglycemic | -3.065 [-16.507 to 10.376] | -4.473 [-18.904 to 9.958] | 2.579 [-8.102 to 13.259] | 2.128 [-8.426 to 12.681] | -3.994 [-14.722 to 6.735]
  T2DM: number analyzed (Participants) | 11 | 10 | 15 | 17 | 15
  T2DM | 3.727 [-6.379 to 13.833] | -1.562 [-12.127 to 9.004] | -1.295 [-10.099 to 7.510] | 6.803 [-1.311 to 14.917] | 2.942 [-5.699 to 11.584]
Statistical Analysis 1: Comparison: LIK066 2.5mg qd vs Placebo; Overall Study; Test type: Other — Dose Finding; p = 0.802, ANCOVA; Mean Difference (Final Values) = 1.308, 95% CI 2-sided [-9.001 to 11.617], Standard Error of Mean 5.2049
Statistical Analysis 2: Comparison: LIK066 10mg qd vs Placebo; Overall Study; Test type: Other — Dose Finding; p = 0.739, ANCOVA; Mean Difference (Final Values) = -1.812, 95% CI 2-sided [-12.567 to 8.943], Standard Error of Mean 5.4301
Statistical Analysis 3: Comparison: LIK066 25 mg qd vs Placebo; Overall Study; Test type: Other — Dose Finding; p = 0.901, ANCOVA; Mean Difference (Final Values) = 0.588, 95% CI 2-sided [-8.745 to 9.922], Standard Error of Mean 4.7125
Statistical Analysis 4: Comparison: LIK066 50 mg qd vs Placebo; Overall Study; Test type: Other — Dose Finding; p = 0.255, ANCOVA; Mean Difference (Final Values) = 5.278, 95% CI 2-sided [-3.852 to 14.407], Standard Error of Mean 4.6095
Statistical Analysis 5: Comparison: LIK066 2.5mg qd vs Placebo; Dysglycemic; Test type: Other — Dose Finding; p = 0.914, ANCOVA; Mean Difference (Final Values) = 0.928, 95% CI 2-sided [-16.271 to 18.127], Standard Error of Mean 8.5585
Statistical Analysis 6: Comparison: LIK066 10mg qd vs Placebo; Dysglycemic; Test type: Other — Dose Finding; p = 0.959, ANCOVA; Mean Difference (Final Values) = -0.480, 95% CI 2-sided [-19.030 to 18.070], Standard Error of Mean 9.2308
Statistical Analysis 7: Comparison: LIK066 25 mg qd vs Placebo; Dysglycemic; Test type: Other — Dose Finding; p = 0.380, ANCOVA; Mean Difference (Final Values) = 6.572, 95% CI 2-sided [-8.343 to 21.487], Standard Error of Mean 7.4220
Statistical Analysis 8: Comparison: LIK066 50 mg qd vs Placebo; Dysglycemic; Test type: Other — Dose Finding; p = 0.419, ANCOVA; Mean Difference (Final Values) = 6.121, 95% CI 2-sided [-8.986 to 21.228], Standard Error of Mean 7.5174
Statistical Analysis 9: Comparison: LIK066 2.5mg qd vs Placebo; T2DM; Test type: Other — Dose Finding; p = 0.906, ANCOVA; Mean Difference (Final Values) = 0.785, 95% CI 2-sided [-12.450 to 14.020], Standard Error of Mean 6.6209
Statistical Analysis 10: Comparison: LIK066 10mg qd vs Placebo; T2DM; Test type: Other — Dose Finding; p = 0.513, ANCOVA; Mean Difference (Final Values) = -4.504, 95% CI 2-sided [-18.195 to 9.187], Standard Error of Mean 6.8489
Statistical Analysis 11: Comparison: LIK066 25 mg qd vs Placebo; T2DM; Test type: Other — Dose Finding; p = 0.499, ANCOVA; Mean Difference (Final Values) = -4.237, 95% CI 2-sided [-16.691 to 8.216], Standard Error of Mean 6.2300
Statistical Analysis 12: Comparison: LIK066 50 mg qd vs Placebo; T2DM; Test type: Other — Dose Finding; p = 0.516, ANCOVA; Mean Difference (Final Values) = 3.860, 95% CI 2-sided [-7.948 to 15.669], Standard Error of Mean 5.9073

13. Secondary Outcome: Percent Change From Baseline at Week 12 on High Sensitive C-reactive Protein (hsCRP)
Description: High sensitivity CRP will be measured from a blood sample and analyzed at a central laboratory. For the overall population and each of the subgroups (Dysglycemic and Type 2 Diabetes Mellitis (T2DM)) from Baseline to Week 12
Time Frame: Baseline, Week 12
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: Percentage
Arm/Group | LIK066 2.5mg qd | LIK066 10mg qd | LIK066 25 mg qd | LIK066 50 mg qd | Placebo
Number analyzed (Participants) | 19 | 19 | 28 | 31 | 29
Percentage
  Overall Study: number analyzed (Participants) | 16 | 16 | 27 | 29 | 28
  Overall Study | -48.448 [-193.256 to 96.359] | 69.004 [-75.849 to 213.858] | -24.207 [-135.765 to 87.352] | -55.536 [-163.215 to 52.144] | -93.268 [-202.833 to 16.296]
  Dysglycemic: number analyzed (Participants) | 7 | 7 | 13 | 13 | 13
  Dysglycemic | 16.582 [-128.374 to 161.538] | 6.593 [-132.996 to 146.182] | -36.745 [-140.259 to 66.770] | -43.562 [-145.987 to 58.864] | -6.298 [-108.747 to 96.151]
  T2DM: number analyzed (Participants) | 9 | 9 | 14 | 16 | 15
  T2DM | -89.337 [-336.322 to 157.648] | 113.169 [-128.460 to 354.798] | -18.143 [-211.748 to 175.463] | -71.025 [-252.712 to 110.662] | -174.159 [-362.344 to 14.026]
Statistical Analysis 1: Comparison: LIK066 2.5mg qd vs Placebo; Overall Study; Test type: Other — Dose Finding; p = 0.625, ANCOVA; Mean Difference (Final Values) = 44.820, 95% CI 2-sided [-136.644 to 226.284]
Statistical Analysis 2: Comparison: LIK066 10mg qd vs Placebo; Overall Study; Test type: Other — Dose Finding; p = 0.079, ANCOVA; Mean Difference (Final Values) = 162.273, 95% CI 2-sided [-19.326 to 343.871]
Statistical Analysis 3: Comparison: LIK066 25 mg qd vs Placebo; Overall Study; Test type: Other — Dose Finding; p = 0.384, ANCOVA; Mean Difference (Final Values) = 69.062, 95% CI 2-sided [-87.493 to 225.617]
Statistical Analysis 4: Comparison: LIK066 50 mg qd vs Placebo; Overall Study; Test type: Other — Dose Finding; p = 0.627, ANCOVA; Mean Difference (Final Values) = 37.733, 95% CI 2-sided [-115.580 to 191.045]
Statistical Analysis 5: Comparison: LIK066 2.5mg qd vs Placebo; Dysglycemic; Test type: Other — Dose Finding; p = 0.797, ANCOVA; Mean Difference (Final Values) = 22.879, 95% CI 2-sided [-155.244 to 201.003]
Statistical Analysis 6: Comparison: LIK066 10mg qd vs Placebo; Dysglycemic; Test type: Other — Dose Finding; p = 0.882, ANCOVA; Mean Difference (Final Values) = 12.891, 95% CI 2-sided [-160.215 to 185.996]
Statistical Analysis 7: Comparison: LIK066 25 mg qd vs Placebo; Dysglycemic; Test type: Other — Dose Finding; p = 0.675, ANCOVA; Mean Difference (Final Values) = -30.447, 95% CI 2-sided [-175.796 to 114.902]
Statistical Analysis 8: Comparison: LIK066 50 mg qd vs Placebo; Dysglycemic; Test type: Other — Dose Finding; p = 0.607, ANCOVA; Mean Difference (Final Values) = -37.264, 95% CI 2-sided [-182.099 to 107.571]
Statistical Analysis 9: Comparison: LIK066 2.5mg qd vs Placebo; T2DM; Test type: Other — Dose Finding; p = 0.591, ANCOVA; Mean Difference (Final Values) = 84.822, 95% CI 2-sided [-229.131 to 398.775]
Statistical Analysis 10: Comparison: LIK066 10mg qd vs Placebo; T2DM; Test type: Other — Dose Finding; p = 0.066, ANCOVA; Mean Difference (Final Values) = 287.328, 95% CI 2-sided [-19.533 to 594.190]
Statistical Analysis 11: Comparison: LIK066 25 mg qd vs Placebo; T2DM; Test type: Other — Dose Finding; p = 0.252, ANCOVA; Mean Difference (Final Values) = 156.017, 95% CI 2-sided [-113.963 to 425.997]
Statistical Analysis 12: Comparison: LIK066 50 mg qd vs Placebo; T2DM; Test type: Other — Dose Finding; p = 0.431, ANCOVA; Mean Difference (Final Values) = 103.135, 95% CI 2-sided [-157.287 to 363.556]

14. Secondary Outcome: Change From Baseline in Uric Acid at Week 12
Description: Uric acid will be measured from a blood sample and analyzed at a central laboratory. For the overall population and each of the subgroups (Dysglycemic and Type 2 Diabetes Mellitis (T2DM)) from Baseline to Week 12
Time Frame: Baseline, Week 12
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: μmol/L
Arm/Group | LIK066 2.5mg qd | LIK066 10mg qd | LIK066 25 mg qd | LIK066 50 mg qd | Placebo
Number analyzed (Participants) | 19 | 19 | 28 | 31 | 29
μmol/L
  Overall Study: number analyzed (Participants) | 19 | 18 | 28 | 30 | 28
  Overall Study | -52.6 [-72.632 to -32.593] | -55.2 [-75.682 to -34.817] | -58.4 [-74.803 to -41.984] | -62.0 [-77.864 to -46.067] | 12.4 [-3.832 to 28.722]
  Dysglycemic: number analyzed (Participants) | 8 | 8 | 13 | 13 | 13
  Dysglycemic | -74.9 [-113.538 to -36.208] | -74.0 [-111.662 to -36.430] | -69.1 [-99.317 to -38.888] | -72.9 [-103.215 to -42.510] | 12.0 [-17.580 to 41.628]
  T2DM: number analyzed (Participants) | 11 | 10 | 15 | 17 | 15
  T2DM | -34.1 [-54.663 to -13.537] | -39.7 [-61.360 to -18.050] | -48.4 [-65.970 to -30.840] | -51.6 [-68.270 to -34.980] | 13.4 [-4.200 to 30.954]
Statistical Analysis 1: Comparison: LIK066 2.5mg qd vs Placebo; Overall Study; Test type: Other — Dose Finding; p < 0.001, ANCOVA; Mean Difference (Final Values) = -65.1, 95% CI 2-sided [-90.864 to -39.251], Standard Error of Mean 13.03
Statistical Analysis 2: Comparison: LIK066 10mg qd vs Placebo; Overall Study; Test type: Other — Dose Finding; p < 0.001, ANCOVA; Mean Difference (Final Values) = -67.7, 95% CI 2-sided [-93.848 to -41.542], Standard Error of Mean 13.21
Statistical Analysis 3: Comparison: LIK066 25 mg qd vs Placebo; Overall Study; Test type: Other — Dose Finding; p < 0.001, ANCOVA; Mean Difference (Final Values) = -70.8, 95% CI 2-sided [-93.942 to -47.735], Standard Error of Mean 11.67
Statistical Analysis 4: Comparison: LIK066 50 mg qd vs Placebo; Overall Study; Test type: Other — Dose Finding; p < 0.001, ANCOVA; Mean Difference (Final Values) = -74.4, 95% CI 2-sided [-97.117 to -51.704], Standard Error of Mean 11.47
Statistical Analysis 5: Comparison: LIK066 2.5mg qd vs Placebo; Dysglycemic; Test type: Other — Dose Finding; p < 0.001, ANCOVA; Mean Difference (Final Values) = -86.9, 95% CI 2-sided [-135.780 to -38.013], Standard Error of Mean 24.35
Statistical Analysis 6: Comparison: LIK066 10mg qd vs Placebo; Dysglycemic; Test type: Other — Dose Finding; p < 0.001, ANCOVA; Mean Difference (Final Values) = -86.1, 95% CI 2-sided [-134.266 to -37.874], Standard Error of Mean 24.01
Statistical Analysis 7: Comparison: LIK066 25 mg qd vs Placebo; Dysglycemic; Test type: Other — Dose Finding; p < 0.001, ANCOVA; Mean Difference (Final Values) = -81.1, 95% CI 2-sided [-123.369 to -38.883], Standard Error of Mean 21.04
Statistical Analysis 8: Comparison: LIK066 50 mg qd vs Placebo; Dysglycemic; Test type: Other — Dose Finding; p < 0.001, ANCOVA; Mean Difference (Final Values) = -84.9, 95% CI 2-sided [-127.104 to -42.669], Standard Error of Mean 21.03
Statistical Analysis 9: Comparison: LIK066 2.5mg qd vs Placebo; T2DM; Test type: Other — Dose Finding; p < 0.001, ANCOVA; Mean Difference (Final Values) = -47.5, 95% CI 2-sided [-74.493 to -20.461], Standard Error of Mean 13.52
Statistical Analysis 10: Comparison: LIK066 10mg qd vs Placebo; T2DM; Test type: Other — Dose Finding; p < 0.001, ANCOVA; Mean Difference (Final Values) = -53.1, 95% CI 2-sided [-80.914 to -25.251], Standard Error of Mean 13.93
Statistical Analysis 11: Comparison: LIK066 25 mg qd vs Placebo; T2DM; Test type: Other — Dose Finding; p < 0.001, ANCOVA; Mean Difference (Final Values) = -61.8, 95% CI 2-sided [-86.627 to -36.937], Standard Error of Mean 12.43
Statistical Analysis 12: Comparison: LIK066 50 mg qd vs Placebo; T2DM; Test type: Other — Dose Finding; p < 0.001, ANCOVA; Mean Difference (Final Values) = -65.0, 95% CI 2-sided [-89.291 to -40.713], Standard Error of Mean 12.15

15. Secondary Outcome: Change From Baseline on Urine Albumin at Week 12
Description: Urine albumin will be measured from urine sample and analyzed at a central laboratory. For the overall population and each of the subgroups (Dysglycemic and Type 2 Diabetes Mellitis (T2DM)) from Baseline to Week 12
Time Frame: Baseline, Week 12
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: x 10^4 mmol/L
Arm/Group | LIK066 2.5mg qd | LIK066 10mg qd | LIK066 25 mg qd | LIK066 50 mg qd | Placebo
Number analyzed (Participants) | 19 | 19 | 28 | 31 | 29
x 10^4 mmol/L
  Overall Study: number analyzed (Participants) | 19 | 18 | 28 | 30 | 28
  Overall Study | -1.838 [-4.665 to 0.990] | 0.008 [-2.891 to 2.907] | -3.902 [-6.233 to -1.572] | -3.099 [-5.360 to -0.838] | -1.282 [-3.603 to 1.040]
  Dysglycemic: number analyzed (Participants) | 8 | 8 | 13 | 13 | 13
  Dysglycemic | -1.941 [-3.792 to -0.089] | 2.030 [0.184 to 3.875] | -2.456 [-3.934 to -0.978] | -3.406 [-4.857 to -1.954] | -3.611 [-5.062 to -2.161]
  T2DM: number analyzed (Participants) | 11 | 10 | 15 | 17 | 15
  T2DM | -3.899 [-7.776 to -0.022] | -1.051 [-5.051 to 2.949] | -3.605 [-6.864 to -0.345] | -2.165 [-5.262 to 0.932] | -0.174 [-3.442 to 3.094]
Statistical Analysis 1: Comparison: LIK066 2.5mg qd vs Placebo; Overall Study; Test type: Other — Dose Finding; p = 0.764, ANCOVA; Mean Difference (Final Values) = -0.556, 95% CI 2-sided [-4.210 to 3.098], Standard Error of Mean 1.8450
Statistical Analysis 2: Comparison: LIK066 10mg qd vs Placebo; Overall Study; Test type: Other — Dose Finding; p = 0.493, ANCOVA; Mean Difference (Final Values) = 1.289, 95% CI 2-sided [-2.423 to 5.001], Standard Error of Mean 1.8741
Statistical Analysis 3: Comparison: LIK066 25 mg qd vs Placebo; Overall Study; Test type: Other — Dose Finding; p = 0.117, ANCOVA; Mean Difference (Final Values) = -2.621, 95% CI 2-sided [-5.908 to 0.666], Standard Error of Mean 1.6596
Statistical Analysis 4: Comparison: LIK066 50 mg qd vs Placebo; Overall Study; Test type: Other — Dose Finding; p = 0.269, ANCOVA; Mean Difference (Final Values) = -1.818, 95% CI 2-sided [-5.056 to 1.421], Standard Error of Mean 1.6349
Statistical Analysis 5: Comparison: LIK066 2.5mg qd vs Placebo; Dysglycemic; Test type: Other — Dose Finding; p = 0.159, ANCOVA; Mean Difference (Final Values) = 1.671, 95% CI 2-sided [-0.676 to 4.017], Standard Error of Mean 1.1677
Statistical Analysis 6: Comparison: LIK066 10mg qd vs Placebo; Dysglycemic; Test type: Other — Dose Finding; p < 0.001, ANCOVA; Mean Difference (Final Values) = 5.641, 95% CI 2-sided [3.294 to 7.988], Standard Error of Mean 1.1678
Statistical Analysis 7: Comparison: LIK066 25 mg qd vs Placebo; Dysglycemic; Test type: Other — Dose Finding; p = 0.271, ANCOVA; Mean Difference (Final Values) = 1.155, 95% CI 2-sided [-0.929 to 3.239], Standard Error of Mean 1.0371
Statistical Analysis 8: Comparison: LIK066 50 mg qd vs Placebo; Dysglycemic; Test type: Other — Dose Finding; p = 0.841, ANCOVA; Mean Difference (Final Values) = 0.206, 95% CI 2-sided [-1.842 to 2.253], Standard Error of Mean 1.0190
Statistical Analysis 9: Comparison: LIK066 2.5mg qd vs Placebo; T2DM; Test type: Other — Dose Finding; p = 0.144, ANCOVA; Mean Difference (Final Values) = -3.725, 95% CI 2-sided [-8.758 to 1.309], Standard Error of Mean 2.5180
Statistical Analysis 10: Comparison: LIK066 10mg qd vs Placebo; T2DM; Test type: Other — Dose Finding; p = 0.736, ANCOVA; Mean Difference (Final Values) = -0.877, 95% CI 2-sided [-6.055 to 4.302], Standard Error of Mean 2.5906
Statistical Analysis 11: Comparison: LIK066 25 mg qd vs Placebo; T2DM; Test type: Other — Dose Finding; p = 0.143, ANCOVA; Mean Difference (Final Values) = -3.431, 95% CI 2-sided [-8.051 to 1.190], Standard Error of Mean 2.3113
Statistical Analysis 12: Comparison: LIK066 50 mg qd vs Placebo; T2DM; Test type: Other — Dose Finding; p = 0.383, ANCOVA; Mean Difference (Final Values) = -1.991, 95% CI 2-sided [-6.521 to 2.538], Standard Error of Mean 2.2659

16. Secondary Outcome: Change From Baseline on Urine Albumin to Creatinine Ratio at Week 12
Description: Urine albumin to creatinine ratio will be measured from urine sample and analyzed at a central laboratory. For the overall population and each of the subgroups (Dysglycemic and Type 2 Diabetes Mellitis (T2DM)) from Baseline to Week 12
Time Frame: Baseline, Week 12
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: mg/mmol
Arm/Group | LIK066 2.5mg qd | LIK066 10mg qd | LIK066 25 mg qd | LIK066 50 mg qd | Placebo
Number analyzed (Participants) | 19 | 19 | 28 | 31 | 29
mg/mmol
  Overall Study: number analyzed (Participants) | 19 | 18 | 27 | 30 | 27
  Overall Study | -0.849 [-2.602 to 0.903] | -0.848 [-2.648 to 0.951] | -2.552 [-4.021 to -1.083] | -1.878 [-3.283 to -0.473] | -1.504 [-2.975 to -0.032]
  Dysglycemic: number analyzed (Participants) | 8 | 8 | 13 | 13 | 13
  Dysglycemic | -0.553 [-1.449 to 0.343] | 0.487 [-0.411 to 1.384] | -0.771 [-1.481 to -0.061] | -1.018 [-1.718 to -0.319] | -1.122 [-1.826 to -0.419]
  T2DM: number analyzed (Participants) | 11 | 10 | 14 | 17 | 14
  T2DM | -1.234 [-4.334 to 1.867] | -1.863 [-5.117 to 1.391] | -4.005 [-6.751 to -1.259] | -2.631 [-5.146 to -0.116] | -1.839 [-4.612 to 0.934]
Statistical Analysis 1: Comparison: LIK066 2.5mg qd vs Placebo; Overall Study; Test type: Other — Dose Finding; p = 0.572, ANCOVA; Mean Difference (Final Values) = 0.654, 95% CI 2-sided [-1.632 to 2.941], Standard Error of Mean 1.1543
Statistical Analysis 2: Comparison: LIK066 10mg qd vs Placebo; Overall Study; Test type: Other — Dose Finding; p = 0.578, ANCOVA; Mean Difference (Final Values) = 0.655, 95% CI 2-sided [-1.670 to 2.980], Standard Error of Mean 1.1738
Statistical Analysis 3: Comparison: LIK066 25 mg qd vs Placebo; Overall Study; Test type: Other — Dose Finding; p = 0.319, ANCOVA; Mean Difference (Final Values) = -1.048, 95% CI 2-sided [-3.124 to 1.028], Standard Error of Mean 1.0479
Statistical Analysis 4: Comparison: LIK066 50 mg qd vs Placebo; Overall Study; Test type: Other — Dose Finding; p = 0.717, ANCOVA; Mean Difference (Final Values) = -0.374, 95% CI 2-sided [-2.416 to 1.667], Standard Error of Mean 1.0303
Statistical Analysis 5: Comparison: LIK066 2.5mg qd vs Placebo; Dysglycemic; Test type: Other — Dose Finding; p = 0.317, ANCOVA; Mean Difference (Final Values) = 0.570, 95% CI 2-sided [-0.562 to 1.701], Standard Error of Mean 0.5630
Statistical Analysis 6: Comparison: LIK066 10mg qd vs Placebo; Dysglycemic; Test type: Other — Dose Finding; p = 0.007, ANCOVA; Mean Difference (Final Values) = 1.609, 95% CI 2-sided [0.460 to 2.758], Standard Error of Mean 0.5716
Statistical Analysis 7: Comparison: LIK066 25 mg qd vs Placebo; Dysglycemic; Test type: Other — Dose Finding; p = 0.487, ANCOVA; Mean Difference (Final Values) = 0.352, 95% CI 2-sided [-0.659 to 1.362], Standard Error of Mean 0.5029
Statistical Analysis 8: Comparison: LIK066 50 mg qd vs Placebo; Dysglycemic; Test type: Other — Dose Finding; p = 0.833, ANCOVA; Mean Difference (Final Values) = 0.104, 95% CI 2-sided [-0.884 to 1.092], Standard Error of Mean 0.4917
Statistical Analysis 9: Comparison: LIK066 2.5mg qd vs Placebo; T2DM; Test type: Other — Dose Finding; p = 0.771, ANCOVA; Mean Difference (Final Values) = 0.605, 95% CI 2-sided [-3.541 to 4.752], Standard Error of Mean 2.0730
Statistical Analysis 10: Comparison: LIK066 10mg qd vs Placebo; T2DM; Test type: Other — Dose Finding; p = 0.991, ANCOVA; Mean Difference (Final Values) = -0.024, 95% CI 2-sided [-4.315 to 4.267], Standard Error of Mean 2.1453
Statistical Analysis 11: Comparison: LIK066 25 mg qd vs Placebo; T2DM; Test type: Other — Dose Finding; p = 0.271, ANCOVA; Mean Difference (Final Values) = -2.166, 95% CI 2-sided [-6.064 to 1.732], Standard Error of Mean 1.9486
Statistical Analysis 12: Comparison: LIK066 50 mg qd vs Placebo; T2DM; Test type: Other — Dose Finding; p = 0.676, ANCOVA; Mean Difference (Final Values) = -0.792, 95% CI 2-sided [-4.570 to 2.986], Standard Error of Mean 1.8889

17. Secondary Outcome: Percent Change From Baseline on Visceral Fat Area (VFA) at Week 12
Description: VFA by CT scan will be measured at visits and evaluated centrally. For the overall population and each of the subgroups (Dysglycemic and Type 2 Diabetes Mellitis (T2DM)) from Baseline to Week 12
Time Frame: Baseline, Week 12
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: Percent
Arm/Group | LIK066 2.5mg qd | LIK066 10mg qd | LIK066 25 mg qd | LIK066 50 mg qd | Placebo
Number analyzed (Participants) | 19 | 19 | 28 | 31 | 29
Percent
  Overall Study | -4.139 [-11.464 to 3.185] | -5.832 [-13.164 to 1.500] | -9.185 [-15.209 to -3.161] | -11.352 [-17.098 to -5.606] | -3.949 [-9.865 to 1.967]
  Dysglycemic: number analyzed (Participants) | 8 | 9 | 13 | 13 | 14
  Dysglycemic | -1.532 [-11.150 to 8.085] | -6.438 [-15.501 to 2.625] | -5.977 [-13.567 to 1.612] | -7.333 [-14.876 to 0.209] | -0.390 [-7.673 to 6.893]
  T2DM: number analyzed (Participants) | 11 | 10 | 15 | 18 | 15
  T2DM | -6.461 [-17.485 to 4.563] | -5.934 [-17.568 to 5.699] | -12.916 [-22.387 to -3.445] | -14.728 [-23.368 to -6.087] | -7.137 [-16.553 to 2.280]
Statistical Analysis 1: Comparison: LIK066 2.5mg qd vs Placebo; Overall Study; Test type: Other — Dose Finding; p = 0.968, ANCOVA; Mean Difference (Final Values) = -0.190, 95% CI 2-sided [-9.603 to 9.222], Standard Error of Mean 4.7535
Statistical Analysis 2: Comparison: LIK066 10mg qd vs Placebo; Overall Study; Test type: Other — Dose Finding; p = 0.693, ANCOVA; Mean Difference (Final Values) = -1.883, 95% CI 2-sided [-11.297 to 7.531], Standard Error of Mean 4.7545
Statistical Analysis 3: Comparison: LIK066 25 mg qd vs Placebo; Overall Study; Test type: Other — Dose Finding; p = 0.222, ANCOVA; Mean Difference (Final Values) = -5.236, 95% CI 2-sided [-13.676 to 3.203], Standard Error of Mean 4.2623
Statistical Analysis 4: Comparison: LIK066 50 mg qd vs Placebo; Overall Study; Test type: Other — Dose Finding; p = 0.078, ANCOVA; Mean Difference (Final Values) = -7.403, 95% CI 2-sided [-15.648 to 0.841], Standard Error of Mean 4.1637
Statistical Analysis 5: Comparison: LIK066 2.5mg qd vs Placebo; Dysglycemic; Test type: Other — Dose Finding; p = 0.850, ANCOVA; Mean Difference (Final Values) = -1.142, 95% CI 2-sided [-13.194 to 10.910], Standard Error of Mean 6.0033
Statistical Analysis 6: Comparison: LIK066 10mg qd vs Placebo; Dysglycemic; Test type: Other — Dose Finding; p = 0.301, ANCOVA; Mean Difference (Final Values) = -6.048, 95% CI 2-sided [-17.676 to 5.580], Standard Error of Mean 5.7919
Statistical Analysis 7: Comparison: LIK066 25 mg qd vs Placebo; Dysglycemic; Test type: Other — Dose Finding; p = 0.293, ANCOVA; Mean Difference (Final Values) = -5.587, 95% CI 2-sided [-16.147 to 4.972], Standard Error of Mean 5.2598
Statistical Analysis 8: Comparison: LIK066 50 mg qd vs Placebo; Dysglycemic; Test type: Other — Dose Finding; p = 0.189, ANCOVA; Mean Difference (Final Values) = -6.943, 95% CI 2-sided [-17.421 to 3.535], Standard Error of Mean 5.2191
Statistical Analysis 9: Comparison: LIK066 2.5mg qd vs Placebo; T2DM; Test type: Other — Dose Finding; p = 0.926, ANCOVA; Mean Difference (Final Values) = 0.676, 95% CI 2-sided [-13.800 to 15.152], Standard Error of Mean 7.2441
Statistical Analysis 10: Comparison: LIK066 10mg qd vs Placebo; T2DM; Test type: Other — Dose Finding; p = 0.873, ANCOVA; Mean Difference (Final Values) = 1.202, 95% CI 2-sided [-13.802 to 16.207], Standard Error of Mean 7.5086
Statistical Analysis 11: Comparison: LIK066 25 mg qd vs Placebo; T2DM; Test type: Other — Dose Finding; p = 0.391, ANCOVA; Mean Difference (Final Values) = -5.779, 95% CI 2-sided [-19.164 to 7.605], Standard Error of Mean 6.6977
Statistical Analysis 12: Comparison: LIK066 50 mg qd vs Placebo; T2DM; Test type: Other — Dose Finding; p = 0.239, ANCOVA; Mean Difference (Final Values) = -7.591, 95% CI 2-sided [-20.345 to 5.163], Standard Error of Mean 6.3822

18. Secondary Outcome: Percent Change From Baseline on Subcutaneous Fat Area (SFA) at Week 12
Description: SFA by CT scan will be measured at visits and evaluated centrally. For the overall population and each of the subgroups (Dysglycemic and Type 2 Diabetes Mellitis (T2DM)) from Baseline to Week 12
Time Frame: Baseline, Week 12
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: Percentage
Arm/Group | LIK066 2.5mg qd | LIK066 10mg qd | LIK066 25 mg qd | LIK066 50 mg qd | Placebo
Number analyzed (Participants) | 19 | 19 | 28 | 31 | 29
Percentage
  Overall Study: number analyzed (Participants) | 19 | 18 | 28 | 31 | 27
  Overall Study | -6.562 [-10.835 to -2.290] | -4.454 [-8.812 to -0.095] | -7.983 [-11.479 to -4.488] | -5.745 [-9.068 to -2.422] | -3.477 [-7.051 to 0.097]
  Dysglycemic: number analyzed (Participants) | 8 | 9 | 13 | 13 | 13
  Dysglycemic | -7.745 [-14.320 to -1.169] | -5.962 [-12.310 to 0.386] | -7.234 [-12.449 to -2.018] | -2.127 [-7.286 to 3.031] | -4.328 [-9.502 to 0.845]
  T2DM: number analyzed (Participants) | 11 | 9 | 15 | 18 | 14
  T2DM | -5.457 [-11.198 to 0.284] | -3.646 [-9.864 to 2.571] | -8.415 [-13.227 to -3.602] | -8.481 [-12.874 to -4.087] | -2.821 [-7.865 to 2.223]
Statistical Analysis 1: Comparison: LIK066 2.5mg qd vs Placebo; Overall Study; Test type: Other — Dose Finding; p = 0.278, ANCOVA; Mean Difference (Final Values) = -3.086, 95% CI 2-sided [-8.696 to 2.525], Standard Error of Mean 2.8326
Statistical Analysis 2: Comparison: LIK066 10mg qd vs Placebo; Overall Study; Test type: Other — Dose Finding; p = 0.733, ANCOVA; Mean Difference (Final Values) = -0.977, 95% CI 2-sided [-6.639 to 4.686], Standard Error of Mean 2.8590
Statistical Analysis 3: Comparison: LIK066 25 mg qd vs Placebo; Overall Study; Test type: Other — Dose Finding; p = 0.075, ANCOVA; Mean Difference (Final Values) = -4.507, 95% CI 2-sided [-9.482 to 0.468], Standard Error of Mean 2.5118
Statistical Analysis 4: Comparison: LIK066 50 mg qd vs Placebo; Overall Study; Test type: Other — Dose Finding; p = 0.360, ANCOVA; Mean Difference (Final Values) = -2.268, 95% CI 2-sided [-7.152 to 2.616], Standard Error of Mean 2.4659
Statistical Analysis 5: Comparison: LIK066 2.5mg qd vs Placebo; Dysglycemic; Test type: Other — Dose Finding; p = 0.416, ANCOVA; Mean Difference (Final Values) = -3.147, 95% CI 2-sided [-11.792 to 4.959], Standard Error of Mean 4.1699
Statistical Analysis 6: Comparison: LIK066 10mg qd vs Placebo; Dysglycemic; Test type: Other — Dose Finding; p = 0.693, ANCOVA; Mean Difference (Final Values) = -1.634, 95% CI 2-sided [-9.893 to 6.625], Standard Error of Mean 4.1121
Statistical Analysis 7: Comparison: LIK066 25 mg qd vs Placebo; Dysglycemic; Test type: Other — Dose Finding; p = 0.428, ANCOVA; Mean Difference (Final Values) = -2.906, 95% CI 2-sided [-10.207 to 4.396], Standard Error of Mean 3.6351
Statistical Analysis 8: Comparison: LIK066 50 mg qd vs Placebo; Dysglycemic; Test type: Other — Dose Finding; p = 0.548, ANCOVA; Mean Difference (Final Values) = 2.201, 95% CI 2-sided [-5.113 to 9.515], Standard Error of Mean 3.6414
Statistical Analysis 9: Comparison: LIK066 2.5mg qd vs Placebo; T2DM; Test type: Other — Dose Finding; p = 0.500, ANCOVA; Mean Difference (Final Values) = -2.636, 95% CI 2-sided [-10.400 to 5.128], Standard Error of Mean 3.8828
Statistical Analysis 10: Comparison: LIK066 10mg qd vs Placebo; T2DM; Test type: Other — Dose Finding; p = 0.837, ANCOVA; Mean Difference (Final Values) = -0.826, 95% CI 2-sided [-8.805 to 7.154], Standard Error of Mean 3.9906
Statistical Analysis 11: Comparison: LIK066 25 mg qd vs Placebo; T2DM; Test type: Other — Dose Finding; p = 0.113, ANCOVA; Mean Difference (Final Values) = -5.594, 95% CI 2-sided [-12.556 to 1.368], Standard Error of Mean 3.4818
Statistical Analysis 12: Comparison: LIK066 50 mg qd vs Placebo; T2DM; Test type: Other — Dose Finding; p = 0.096, ANCOVA; Mean Difference (Final Values) = -5.660, 95% CI 2-sided [-12.361 to 1.041], Standard Error of Mean 3.3512

19. Secondary Outcome: Pharmacokinetics - Plasma Trough Concentrations of LIK066
Description: Plasma trough concentrations of LIK066 were measured at Week 12 after daily administrations of LIK066 (2.5, 10, 25 and 50 mg).
Time Frame: Week 12
Population: Safety set (SAF): the SAF includes all participants who received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | LIK066 2.5mg qd | LIK066 10mg qd | LIK066 25 mg qd | LIK066 50 mg qd
Number analyzed (Participants) | 19 | 19 | 28 | 31
ng/mL | 1.63 (0.947) | 4.17 (2.94) | 12.8 (8.56) | 26.4 (21.8)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected till the end of the study.(about 12 weeks) and serious adverse events (SAEs) were collected until 30 days after the last study visit (12 weeks + 30 days = about 114 days)
Description: AE additional description
Groups:
- LIK066 25mg qd: Eligible patients randomized to this arm will receive LIK066 25 mg orally daily (qd) for 12 weeks.
- LIK066 50mg qd: Eligible patients randomized to this arm will receive LIK066 50 mg orally daily (qd) for 12 weeks.
Arm/Group | LIK066 2.5mg qd | LIK066 10mg qd | LIK066 25mg qd | LIK066 50mg qd | Placebo
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19 | 0/28 | 0/31 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19 | 0/28 | 1/31 | 0/29
Other Adverse Events (participants affected / at risk) | 10/19 | 12/19 | 13/28 | 20/31 | 9/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LIK066 2.5mg qd (N=19) | LIK066 10mg qd (N=19) | LIK066 25mg qd (N=28) | LIK066 50mg qd (N=31) | Placebo (N=29)
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LIK066 2.5mg qd (N=19) | LIK066 10mg qd (N=19) | LIK066 25mg qd (N=28) | LIK066 50mg qd (N=31) | Placebo (N=29)
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 4 | 12 | 2
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0
Gastric polyps (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Gastritis erosive (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Malaise (General disorders) | 0 | 1 | 0 | 0 | 0
Hepatic steatosis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 1
Asymptomatic bacteriuria (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 1 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Gingivitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 2 | 3 | 5 | 4 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0
Protein urine present (Investigations) | 1 | 0 | 2 | 0 | 1
Urine albumin/creatinine ratio increased (Investigations) | 0 | 2 | 0 | 2 | 2
White blood cells urine positive (Investigations) | 1 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 2 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 2
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety

DOCUMENTS (2):
  • Study Protocol (2017-10-30): https://cdn.clinicaltrials.gov/large-docs/41/NCT03320941/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-13): https://cdn.clinicaltrials.gov/large-docs/41/NCT03320941/SAP_001.pdf